CLINICAL TRIAL: NCT06421909
Title: Effect of Mindfulness-based Educational Intervention on Anxiety, Depression, Stress and Quality of Life on Menopausal Woman.
Brief Title: Mindfulness-based Educational Intervention on Anxiety, Depression, Stress and Quality of Life on Menopausal Woman
Acronym: mindmenopaus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 99-b
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based educational intervention group (Experimental)
  Interventions: Behavioral: mindfulness-based educational intervention
- non-intervention group (No Intervention)

INTERVENTIONS:
Behavioral: mindfulness-based educational intervention — Mindfulness-based educational intervention is a structured program that incorporates principles of mindfulness to help individuals develop greater awareness and acceptance of their thoughts, feelings, and bodily sensations. The intervention typically includes mindfulness meditation practices, cognitive-behavioral techniques, and educational components about stress management and emotional regulation. By fostering a non-judgmental and present-focused attitude, participants learn to manage their symptoms more effectively and improve their overall quality of life.
  Arms: mindfulness-based educational intervention group

SUMMARY:
Mindfulness-based educational intervention is a structured program that incorporates principles of mindfulness to help individuals develop greater awareness and acceptance of their thoughts, feelings, and bodily sensations. The intervention typically includes mindfulness meditation practices, cognitive-behavioral techniques, and educational components about stress management and emotional regulation. By fostering a non-judgmental and present-focused attitude, participants learn to manage their symptoms more effectively and improve their overall quality of life.

DETAILED DESCRIPTION:
Menopause is a significant transitional phase in a woman's life, often accompanied by various physical, emotional, and psychological challenges. Common issues during menopause include anxiety, depression, stress, and a decreased quality of life. Addressing these concerns holistically is crucial for improving overall well-being. Mindfulness-based educational interventions have gained recognition for their effectiveness in enhancing mental health and quality of life by promoting awareness and acceptance of present experiences. This study investigates the impact of a mindfulness-based educational intervention on anxiety, depression, stress, and quality of life in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* in age of menopause

Exclusion Criteria:

* age of menarche
* older than 70 years old

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
menopausal women who participate in the mindfulness-based educational intervention will experience significant reductions in anxiety inventory score ( total score range from 10 to 50, a lower score of less than 20) than those who not entered | three months

SECONDARY OUTCOMES:
menopausal women who participate in the mindfulness-based educational intervention will experience reductions in stress scale score ( total score range from 10 to 50, a lower score of less than 20) than those who not entered | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Alexandria Governorate, Egypt

REFERENCES:
- [Derived] Amin SM, El-Gazar HE, Zoromba MA, El-Sayed MM, Awad AGE, Atta MHR. Mindfulness for Menopausal Women: Enhancing Quality of Life and Psychological Well-Being Through a Randomized Controlled Intervention. J Nurs Scholarsh. 2025 Jul;57(4):563-575. doi: 10.1111/jnu.70003. Epub 2025 Feb 24. PMID 39992004